CLINICAL TRIAL: NCT00118534
Title: CSP #519 - Integrating Practice Guidelines for Smoking Cessation Into Mental Health Care for PTSD (SCP)
Brief Title: Integrating Clinical Practice Guidelines for Smoking Cessation Into Mental Health Care for Veterans With Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 519
Record Dates: First submitted 2005-07-01; First posted 2005-07-11 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Mental Health; Stress Disorders, Post-Traumatic; Substance-Related Disorders; Tobacco Use Disorder
Keywords: addictive disorders; clinical trial; cost effectiveness; mental health; military or environmental exposure; multi-site trial; nicotine; nicotine replacement; post traumatic stress; post traumatic stress disorder; psychiatric; psychological; PTSD; smoking cessation; smoking cessation medications; substance abuse
MeSH Terms: conditions — Psychological Well-Being; Stress Disorders, Post-Traumatic; Substance-Related Disorders; Tobacco Use Disorder; Smoking Cessation | interventions — Delivery of Health Care, Integrated; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Integration of smoking cessation therapy with PTSD therapy.
  Interventions: Behavioral: Integrated Care for Smoking Cessation in PTSD patients
- Arm 2 (Active Comparator): Per standard of care, patients are referred to a smoking cessation clinic for their smoking cessation therapy.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Integrated Care for Smoking Cessation in PTSD patients — Smoking cessation therapy is integrated with PTSD therapy.
  Other Names: Integrated Care (IC)
  Arms: Arm 1
Behavioral: Standard of Care — Patients interested in quitting smoking are referred to a separate smoking cessation clinic, per standard of care.
  Arms: Arm 2

SUMMARY:
The primary study objective is to conduct a prospective, randomized controlled clinical trial that compares the effectiveness of two approaches for delivering smoking cessation treatment for veterans with posttraumatic stress disorder (PTSD). An approach where smoking cessation treatment is integrated into mental health care for PTSD and delivered by mental health providers (experimental condition) will be compared to specialized smoking cessation clinic referral (VA's usual standard of care).

Secondary study objectives are to (a) compare the cost outcomes and cost-effectiveness of IC versus USC, (b) identify treatment process variables that explain (mediate) observed differences in smoking abstinence rates for the two study conditions, and (c) determine whether cessation from smoking is associated with worsening of symptoms of PTSD and/or depression.

DETAILED DESCRIPTION:
Intervention: The research will test the effectiveness of integrating evidence-based, efficacious treatments for tobacco use disorder into mental health care for patients with chronic PTSD. Two different methods for delivering smoking cessation treatment will be compared in a randomized, controlled clinical effectiveness trial conducted at four Department of Veterans Affairs (VA) medical centers. Smokers undergoing mental health care for PTSD who want to quit smoking will be randomly assigned to either (1) guideline-concordant smoking cessation treatment integrated within ongoing mental health care for PTSD, and delivered by mental health providers (Integrated Care (IC), experimental condition), or (2) specialized smoking cessation treatment, delivered separately from PTSD treatment by a smoking cessation clinic (Usual Standard of Care (USC), comparison condition).

Primary Hypothesis: IC will be more effective than USC on measures of smoking-related clinical outcomes.

Secondary Hypothesis: The following treatment process variables will predict smoking abstinence at 12-months post randomization: (a) number of smoking cessation treatment sessions received, (b) type and duration of protocol medications prescribed by providers (bupropion, transdermal nicotine patch, and nicotine gum), (c) degree of subjects' compliance with prescribed protocol medication, and (d) number of quit attempts marked by abstinence of 7 days or more.

Treatment process variables that predict smoking abstinence will be present to a significantly greater degree in IC than USC.

Primary Outcomes: The primary outcome measure will be the point-prevalence of smoking abstinence by self-report for the 7 days prior to assessments, obtained at months 3, 6, 9, and 12 following randomization to study conditions. Verification of smoking abstinence will be obtained by CO readings (abstinence < 10 ppm) obtained at each assessment interval. Salivary cotinine levels (abstinence < 20 ng/ml) will be measured to verify abstinence at months 9 and 12 only, as subjects may still be using nicotine replacement medicines at earlier assessment intervals, confounding cotinine assays.

Study Abstract: Individuals with posttraumatic stress disorder (PTSD) are far more likely to smoke than those without mental illness and they smoke more heavily. Tobacco use likely contributes to the heightened overall mortality and specific risks for smoking related diseases among veterans with PTSD and commonly co-occurring mental disorders.

Symptoms of PTSD and associated mental disorders are linked to the maintenance of tobacco dependence, premature dropout from smoking cessation treatment, and relapse to smoking following quit attempts. Many efficacious tobacco use treatments exist, but a number of barriers limit the effectiveness of current methods for delivering these treatments in VA health care settings, particularly for the mentally ill. Novel approaches to smoking cessation for individuals with PTSD are needed to circumvent these barriers by integrating evidence-based tobacco use treatment into ongoing mental health care. The research proposed here will test the effectiveness of integrating evidence-based treatment for nicotine dependence into mental health care for patients with chronic posttraumatic stress disorder (PTSD). Two different methods for delivering smoking cessation treatment will be compared in a prospective, randomized controlled clinical effectiveness trial conducted at four Department of Veterans Affairs (VA) medical centers. Smokers undergoing mental health care for PTSD (n=440) will be randomly assigned to either: (1) practice guideline-concordant smoking cessation treatment that is integrated within ongoing mental health care for PTSD and delivered by mental health providers (Integrated Care [IC]) or 2) smoking cessation treatment delivered separately from PTSD treatment by smoking cessation specialists (Usual Standard of Care [USC]). Specific aims of the proposed investigation are (1) to demonstrate that IC is more effective than USC in reducing smoking in psychiatric patients with PTSD and (2) to demonstrate that a number of treatment process variables, including the amount or dose of intervention and patient-specific factors, predict abstinence from tobacco use in smokers with PTSD. Intent-to-treat analyses and analyses for treatment completers will be conducted, using a Generalized Estimating Equations approach. If the study hypothesis is confirmed, system-wide implementation of the experimental intervention (IC) for veterans with PTSD would double the number of patients who stop smoking compared to the usual standard of care for tobacco use disorder. Study findings may have implications for integrating smoking cessation treatment into mental health care for patients with disorders other than PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Receive a minimum of four mental health treatment sessions from the SOPP that span at least a 1-month interval
* SOPP treatment plan must indicate intent to deliver ongoing PTSD care for at least 1 year, including visits at least once per month
* Diagnosis of PTSD resulting from military trauma using DSM-IV criteria
* Current nicotine use, smoking greater at least 10 cigarettes per day for at least 16 of the past 30 days prior to randomization
* Demonstrated motivation to quit smoking

Exclusion Criteria:

* Use of smokeless tobacco or smoke pipes or cigars
* Any psychotic disorder that is not in remission
* Bipolar disorder that is not in remission
* Any substance dependence disorder that is not in remission (current substance abuse disorder and substance dependence disorder in remission for more than 1 month are not exclusions)
* Imminent risk for suicide or violence, as determined during routine assessment by SOPP clinical staff
* Severe psychiatric symptoms or psychosocial instability likely to prevent participation in the study protocol (i.e., attendance at scheduled sessions, ability to read study materials, and/or ability to comprehend interventions), as determined during routine assessment by SOPP clinical staff
* Gross impairment from organic mental disorder, as determined during routine assessment by SOPP clinical staff

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 943 (Actual)
Dates: Start 2004-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miles E McFall, PhD, Study Chair — VA Puget Sound Health Care System, Seattle
Locations (11):
- United States (11):
  - VA Medical Center, Tuscaloosa, Tuscaloosa, Alabama
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - VA Medical Center, DC, Washington D.C., District of Columbia
  - Southeast Veterans Healthcare System, New Orleans, New Orleans, Louisiana
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Medical Center, Portland, Portland, Oregon
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - VA Medical Center, Providence, Providence, Rhode Island
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - VA Medical Center, Hampton, Hampton, Virginia
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington

REFERENCES:
- [Result] Smith MW, Chen S, Siroka AM, Hamlett-Berry K. Using policy to increase prescribing of smoking cessation medications in the VA healthcare system. Tob Control. 2010 Dec;19(6):507-11. doi: 10.1136/tc.2009.035147. Epub 2010 Sep 24. PMID 20870742
- [Result] McFall M, Saxon AJ, Malte CA, Chow B, Bailey S, Baker DG, Beckham JC, Boardman KD, Carmody TP, Joseph AM, Smith MW, Shih MC, Lu Y, Holodniy M, Lavori PW; CSP 519 Study Team. Integrating tobacco cessation into mental health care for posttraumatic stress disorder: a randomized controlled trial. JAMA. 2010 Dec 8;304(22):2485-93. doi: 10.1001/jama.2010.1769. PMID 21139110
- [Derived] Barnett PG, Jeffers A, Smith MW, Chow BK, McFall M, Saxon AJ. Cost-Effectiveness of Integrating Tobacco Cessation Into Post-Traumatic Stress Disorder Treatment. Nicotine Tob Res. 2016 Mar;18(3):267-74. doi: 10.1093/ntr/ntv094. Epub 2015 May 4. PMID 25943761
- [Derived] Joseph AM, McFall M, Saxon AJ, Chow BK, Leskela J, Dieperink ME, Carmody TP, Beckham JC. Smoking intensity and severity of specific symptom clusters in posttraumatic stress disorder. J Trauma Stress. 2012 Feb;25(1):10-6. doi: 10.1002/jts.21670. Epub 2012 Feb 10. PMID 22328334
- [Derived] Harder LH, Chen S, Baker DG, Chow B, McFall M, Saxon A, Smith MW. The influence of posttraumatic stress disorder numbing and hyperarousal symptom clusters in the prediction of physical health status in veterans with chronic tobacco dependence and posttraumatic stress disorder. J Nerv Ment Dis. 2011 Dec;199(12):940-5. doi: 10.1097/NMD.0b013e3182392bfb. PMID 22134452

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between November 2004 and December 2007, with follow-up continuing until July 2009.943 patients were recruited from outpatient PTSD clinics at 10 VA medical centers and followed up for a minimum of 18 months.
Pre-assignment Details: Patients gave written informed consent before enrollment.
Groups:
- Integrated Care: Integration of smoking cessation therapy with PTSD therapy.
- Standard of Care: Per standard of care, patients are referred to a smoking cessation clinic for their smoking cessation therapy.
Period: Overall Study
Arm/Group | Integrated Care | Standard of Care
Started | 472 | 471
Completed | 472 | 471
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Care | Standard of Care | Total
Number analyzed (Participants) | 472 | 471 | 943
Age, Continuous [Mean (Full Range); unit: years] | 54.4 [22 to 80] | 54.7 [23 to 81] | 54.56 [22 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 60
  Male | 444 | 439 | 883
Region of Enrollment [Number; unit: participants]
  United States | 472 | 471 | 943

OUTCOME MEASURES:

1. Primary Outcome: Bioverified 12-Month Prolonged Abstinence Between 6 and 18 Months Postrandomization
Description: The primary outcome measure was 12-month bio-verified prolonged abstinence from tobacco between 6 and 18 months postrandomization. Prolonged abstinence excluded tobacco use before 6 months postrandomization. Prolonged abstinence defined non-abstinence as 1) smoking for 7 consecutive days or at least once a week for 2 consecutive weeks, or 2) using non-cigarette tobacco for 7 consecutive days or at least once a week for 2 consecutive weeks. Self-reported prolonged abstinence was verified by exhaled CO ≤ 8ppm and urine cotinine <100 ng/mL cotinine equivalents at the 9-18 month visits. If CO or cotinine was missing, a single measure was used for verification. If both CO and cotinine were missing at any visit between 9 and 15 months, patients reporting prolonged abstinence were considered abstinent if all other available bioverification data confirmed abstinence. Patients who lacked CO and cotinine readings at 18 months or failed to attend the 18 month visit were considered nonabstinent.
Time Frame: between 6 and 18 months
Measure: Number; unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 42 | 21
Statistical Analysis 1: Comparison: Integrated Care vs Standard of Care; The target sample size (n=1400)was designed to have 90% power to detect the difference between 6% and 11% prolonged abstinence rates in SCC and IC, respectively, using a 2-sided .05 level Chi-square test. Final enrollment was 943. The recruitment period was not extended because the achieved sample size provided 78% power to detect the hypothesized prolonged abstinence rates, and the study continued to the end of planned follow-up; Test type: Superiority or Other; p = 0.007, Regression, Logistic; Odds Ratio (OR) = 2.09, 95% CI 2-sided [1.22 to 3.59]

2. Secondary Outcome: Self-reported 12-month Prolonged Abstinence Between 6 and 18 Months
Description: A secondary outcome was self-reported 1-year prolonged abstinence between 6 and 18 months post-randomization. Prolonged abstinence excluded tobacco use prior to 6 months post-randomization to allow for initial treatment episode completion and recovery from early relapses. Prolonged abstinence defined non-abstinence as: 1) smoking for 7 consecutive days or at least once a week for 2 consecutive weeks, or 2) using non-cigarette tobacco for 7 consecutive days or at least once a week for 2 consecutive weeks.
Time Frame: between 6 and 18 months
Measure: Number; unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 73 | 33
Statistical Analysis 1: Comparison: Integrated Care vs Standard of Care; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.43, 95% CI 2-sided [1.58 to 3.74]

3. Secondary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: Severity of PTSD was a predetermined secondary outcome. One of the measurements for this was CAPS at 18 months. The range is 0-136; five rationally derived severity score ranges for interpreting CAPS total score have been proposed and are as follows: 0-19 = asymptomatic/few symptoms, 20-39 = mild PTSD/subthreshold, 40-59 = moderate PTSD/threshold, 60-79 = severe PTSD symptomatology, and >80 = extreme PTSD symptomology. A rationally derived 15-point change in CAPS total severity score has been proposed as a marker of clinically significant change. The above severity ranges and 15-point marker are preliminary (Frank W. Weathers et. al., "Clinician-administered PTSD Scale: A Review of the First Ten Years of Research", Depression and Anxiety 13: 132-156 (2001)). The results are reported in mean change from baseline.
Time Frame: Baseline and 18 months
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
Units on a scale | -7.2 [-9.1 to -5.2] | -7.0 [-9.0 to -5.0]

4. Secondary Outcome: PTSD Checklist
Description: Severity of PTSD was a predetermined secondary outcome. One of the measurements for this was PTSD Checklist (range, 17-85; scores of greater or equal to 50 indicate a PTSD diagnosis) at every assessment. The results are reported as the mean change from baseline for the 3 month assessment.
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
units on a scale | -2.0 [-3.0 to -1.0] | -0.9 [-1.9 to 0.2]

5. Secondary Outcome: PTSD Checklist
Description: Severity of PTSD was a predetermined secondary outcome. One of the measurements for this was PTSD Checklist (range, 17-85; scores of greater or equal to 50 indicate a PTSD diagnosis) at every assessment. The results are reported as the mean change from baseline for the 6 month assessment.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
units on a scale | 1.6 [0.5 to 2.7] | 2.2 [1.1 to 3.3]

6. Secondary Outcome: PTSD Checklist
Description: Severity of PTSD was a predetermined secondary outcome. One of the measurements for this was PTSD Checklist (range, 17-85; scores of greater or equal to 50 indicate a PTSD diagnosis) at every assessment. The results are reported as the mean change from baseline for the 9 month assessment.
Time Frame: Baseline and 9 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
units on a scale | -1.4 [-2.5 to -0.4] | -0.9 [-2.0 to 0.2]

7. Secondary Outcome: PTSD Checklist
Description: Severity of PTSD was a predetermined secondary outcome. One of the measurements for this was PTSD Checklist (range, 17-85; scores of greater or equal to 50 indicate a PTSD diagnosis) at every assessment. The results are reported as the mean change from baseline for the 12 month assessment.
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
units on a scale | -1.6 [-2.7 to -0.5] | -1.4 [-2.5 to -0.3]

8. Secondary Outcome: PTSD Checklist
Description: Severity of PTSD was a predetermined secondary outcome. One of the measurements for this was PTSD Checklist (range, 17-85; scores of greater or equal to 50 indicate a PTSD diagnosis) at every assessment. The results are reported as the mean change from baseline for the 15 month assessment.
Time Frame: Baseline and 15 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
units on a scale | -1.8 [-2.9 to -0.8] | -0.9 [-2.0 to 0.2]

9. Secondary Outcome: PTSD Checklist
Description: Severity of PTSD was a predetermined secondary outcome. One of the measurements for this was PTSD Checklist (range, 17-85; scores of greater or equal to 50 indicate a PTSD diagnosis) at every assessment. The results are reported as the mean change from baseline for the 18 month assessment.
Time Frame: Baseline and 18 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
units on a scale | -3.2 [-4.3 to -2.1] | -2.4 [-3.5 to -1.2]

10. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: The Patient Health Questionnaire 9 (PHQ-9; range, 0-27; scores of 10-14, 15-19, and greater than or equal to 20 indicate mild, moderate, and severe depression,respectively) measured depression at every assessment. The results are reported as the mean change from baseline for the 3 month assessment.
Time Frame: Baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
units on a scale | 0.6 [0.1 to 1.0] | 0.9 [0.4 to 1.4]

11. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: The Patient Health Questionnaire 9 (PHQ-9; range, 0-27; scores of 10-14, 15-19, and greater than or equal to 20 indicate mild, moderate, and severe depression,respectively) measured depression at every assessment. The results are reported as the mean change from baseline for the 6 month assessment.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
units on a scale | 0.9 [0.3 to 1.4] | 1.0 [0.4 to 1.5]

12. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: The Patient Health Questionnaire 9 (PHQ-9; range, 0-27; scores of 10-14, 15-19, and greater than or equal to 20 indicate mild, moderate, and severe depression,respectively) measured depression at every assessment. The results are reported as the mean change from baseline for the 9 month assessment.
Time Frame: Baseline and 9 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
units on a scale | 1.1 [0.6 to 1.7] | 1.3 [0.7 to 1.9]

13. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: The Patient Health Questionnaire 9 (PHQ-9; range, 0-27; scores of 10-14, 15-19, and greater than or equal to 20 indicate mild, moderate, and severe depression,respectively) measured depression at every assessment. The results are reported as the mean change from baseline for the 12 month assessment.
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
units on a scale | 1.6 [1.0 to 2.1] | 1.2 [0.6 to 1.8]

14. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire 9 (PHQ-9; range, 0-27; scores of 10-14, 15-19, and greater than or equal to 20 indicate mild, moderate, and severe depression,respectively) measured depression at every assessment. The results are reported as the mean change from baseline for the 15 month assessment.
Time Frame: Baseline and 15 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
units on a scale | 1.1 [0.6 to 1.6] | 1.2 [0.6 to 1.8]

15. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: The Patient Health Questionnaire 9 (PHQ-9; range, 0-27; scores of 10-14, 15-19, and greater than or equal to 20 indicate mild, moderate, and severe depression,respectively) measured depression at every assessment. The results are reported as the mean change from baseline for the 18 month assessment.
Time Frame: Baseline and 18 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
units on a scale | -0.2 [-0.7 to 0.4] | -0.3 [-0.8 to 0.3]

16. Secondary Outcome: 7-day Point Prevalence Abstinence - Self Reported
Description: Predetermined secondary smoking outcomes included 7- and 30-day point prevalence abstinence at each assessment, where abstinence was defined as no tobacco use in the prior 7 or 30 days, respectively. Self-reported point prevalence abstinence was determined for all patients, with patients not completing a visit presumed to be nonabstinent.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 126 [107 to 145] | 65 [50 to 80]

17. Secondary Outcome: 7-day Point Prevalence Abstinence - Self Reported
Description: as for outcome 16
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 132 [113 to 151] | 63 [49 to 77]

18. Secondary Outcome: 7-day Point Prevalence Abstinence - Self Reported
Description: as for outcome 16
Time Frame: 9 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 122 [103 to 141] | 60 [46 to 74]

19. Secondary Outcome: 7-day Point Prevalence Abstinence - Self Reported
Description: as for outcome 16
Time Frame: 12 months
Measure: Number (90% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 117 [99 to 135] | 70 [55 to 85]

20. Secondary Outcome: 7-day Point Prevalence Abstinence - Self Reported
Description: as for outcome 16
Time Frame: 15 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 119 [101 to 137] | 63 [49 to 77]

21. Secondary Outcome: 7-day Point Prevalence Abstinence - Self Reported
Description: as for outcome 16
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 111 [93 to 129] | 73 [58 to 88]

22. Secondary Outcome: 7-day Point Prevalence Abstinence - Bio-Verified
Description: Predetermined secondary smoking outcomes included 7- and 30-day point prevalence abstinence at each assessment, where abstinence was defined as no tobacco use in the prior 7 or 30 days, respectively. Self-reported point prevalence abstinence was determined for all patients, with patients not completing a visit presumed to be nonabstinent. Exhaled carbon monoxide (CO) was obtained at every in person assessment. Urine cotinine levels, using Accutest® NicAlert™ test strips, were ascertained at assessments when patients self-reported no use of tobacco or nicotine replacement therapy in the prior 7 days. Laboratory assays of urine cotinine were obtained when self-reported abstinence disagreed with NicAlert™ results. If bioverification data were missing or did not confirm abstinence, patients were considered nonabstinent at that visit.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 67 [52 to 82] | 37 [26 to 48]

23. Secondary Outcome: 7-day Point Prevalence Abstinence - Bio-Verified
Description: as for outcome 22
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 78 [62 to 94] | 34 [23 to 45]

24. Secondary Outcome: 7-day Point Prevalence Abstinence - Bio-Verified
Description: as for outcome 22
Time Frame: 9 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 70 [55 to 85] | 35 [24 to 46]

25. Secondary Outcome: 7-day Point Prevalence Abstinence - Bio-Verified
Description: as for outcome 22
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 66 [51 to 81] | 44 [32 to 56]

26. Secondary Outcome: 7-day Point Prevalence Abstinence - Bio-Verified
Description: as for outcome 22
Time Frame: 15 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 67 [52 to 82] | 36 [25 to 47]

27. Secondary Outcome: 7-day Point Prevalence Abstinence - Bio-Verified
Description: as for outcome 22
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 86 [70 to 102] | 51 [38 to 64]

28. Secondary Outcome: 30-day Point Prevalence Abstinence - Self Reported
Description: as for outcome 16
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 126 [107 to 145] | 65 [50 to 80]

29. Secondary Outcome: 30-day Point Prevalence Abstinence - Self Reported
Description: as for outcome 16
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 132 [113 to 151] | 63 [49 to 77]

30. Secondary Outcome: 30-day Point Prevalence Abstinence - Self Reported
Description: as for outcome 16
Time Frame: 9 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 122 [103 to 141] | 60 [46 to 74]

31. Secondary Outcome: 30-day Point Prevalence Abstinence - Self Reported
Description: as for outcome 16
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 117 [99 to 135] | 70 [55 to 85]

32. Secondary Outcome: 30-day Point Prevalence Abstinence - Self Reported
Description: as for outcome 16
Time Frame: 15 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 119 [101 to 137] | 63 [49 to 77]

33. Secondary Outcome: 30-day Point Prevalence Abstinence - Self Reported
Description: as for outcome 16
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 111 [93 to 129] | 73 [58 to 88]

34. Secondary Outcome: 30-day Point Prevalence Abstinence - Bio-Verified
Description: as for outcome 22
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 67 [52 to 82] | 37 [26 to 48]

35. Secondary Outcome: 30-day Point Prevalence Abstinence - Bio-Verified
Description: as for outcome 22
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 78 [62 to 94] | 34 [23 to 45]

36. Secondary Outcome: 30-day Point Prevalence Abstinence - Bio-Verified
Description: as for outcome 22
Time Frame: 9 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 70 [55 to 85] | 35 [24 to 46]

37. Secondary Outcome: 30-day Point Prevalence Abstinence - Bio-Verified
Description: as for outcome 22
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 66 [51 to 81] | 44 [32 to 56]

38. Secondary Outcome: 30-day Point Prevalence Abstinence - Bio-Verified
Description: as for outcome 22
Time Frame: 15 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 67 [52 to 82] | 36 [25 to 47]

39. Secondary Outcome: 30-day Point Prevalence Abstinence - Bio-Verified
Description: as for outcome 22
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Integrated Care | Standard of Care
Number analyzed (Participants) | 472 | 471
participants | 86 [70 to 102] | 51 [38 to 64]

ADVERSE EVENTS:
Arm/Group | Integrated Care | Standard of Care
Serious Adverse Events (participants affected / at risk) | 218/472 | 220/471
Other Adverse Events (participants affected / at risk) | 44/472 | 38/471
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Integrated Care (N=472) | Standard of Care (N=471)
Unevaluable event (General disorders) | 8 (9) | 8 (10)
AV nodal reentrant tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Angina attack (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 3 (4) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Congestive cardiac failure aggravated (Cardiac disorders) | 1 (2) | 1 (2)
Congestive heart failure (Cardiac disorders) | 4 (6) | 2 (2)
Constrictive pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 4 (4) | 9 (11)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (2) | 0 (0)
Coronary occlusion (Cardiac disorders) | 1 (2) | 0 (0)
Heart attack (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial infarction (Cardiac disorders) | 8 (10) | 2 (2)
Non STEMI (Cardiac disorders) | 0 (0) | 1 (1)
Non-Q wave MI (Cardiac disorders) | 1 (1) | 0 (0)
Non-ischemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Paroxysmal atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Paroxysmal supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Right heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Unstable angina (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriovenous malformations (Congenital, familial and genetic disorders) | 0 (0) | 1 (2)
Maxillary hypoplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Alternating exotropia (Eye disorders) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Achalasia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Acute pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bleeding duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bleeding gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood in stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Constipation chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
GERD (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI tract bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Left lower quadrant pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Perforated colon (Gastrointestinal disorders) | 0 (0) | 1 (1)
Persistent vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Right inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Uvulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3)
Vomiting blood (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting post chemotherapy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 6 (6) | 8 (9)
Cyst (General disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 2 (2) | 2 (2)
Died in sleep (General disorders) | 1 (1) | 0 (0)
Disease complication (General disorders) | 1 (1) | 0 (0)
Edema (General disorders) | 1 (1) | 0 (0)
Edema of lower extremities (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Opiate withdrawal symptoms (General disorders) | 1 (1) | 0 (0)
Ulcer (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder stones (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Obstructive jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess intestinal (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Abscess on buttock (Infections and infestations) | 1 (1) | 0 (0)
Acute appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Acute bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Asymptomatic neurosyphilis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial meningitis (Infections and infestations) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 3 (3)
Cellulitis of arm (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis of leg (Infections and infestations) | 1 (1) | 2 (3)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Community acquired pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Condyloma (Infections and infestations) | 1 (1) | 0 (0)
Creutzfeldt-Jakob disease (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 4 (5) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Ear infection viral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
HIV infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 2 (2)
Hip osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Infection urinary tract (Infections and infestations) | 0 (0) | 1 (1)
Legionnaire's disease (Infections and infestations) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
MRSA wound infection (Infections and infestations) | 1 (1) | 0 (0)
Methicillin-resistant staphylococcal aureus infection (Infections and infestations) | 0 (0) | 2 (3)
Mouth abscess (Infections and infestations) | 1 (1) | 0 (0)
Nasal abscess (Infections and infestations) | 0 (0) | 1 (1)
Neurosyphilis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 9 (9)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Sialadenitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Spinal osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Surgical wound infection (Infections and infestations) | 1 (1) | 1 (1)
UTI (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Viral gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Viral hepatitis (Infections and infestations) | 0 (0) | 1 (1)
Viral pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Accident at home (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Achilles tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute alcoholic intoxication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol intoxication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Automobile accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Broken leg (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cat bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cataract operation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Collapse of lung (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary stent occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Crushing injury of trunk (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cycling accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Delayed recovery from anesthetic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dumping syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 9 (10)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured ribs (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Implant failure (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Overdose effect (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post biopsy bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural bleeding (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative complication (Injury, poisoning and procedural complications) | 1 (6) | 0 (0)
Postoperative hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rupture tendon (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spider bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sports injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture granuloma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Biopsy larynx normal (Investigations) | 1 (1) | 0 (0)
Blood carbon monoxide increased (Investigations) | 0 (0) | 1 (1)
Blood sugar increased (Investigations) | 1 (1) | 2 (2)
Cardiac catheterization (Investigations) | 1 (1) | 0 (0)
Coronary angiogram (Investigations) | 0 (0) | 1 (1)
Elevated prostate specific antigen [PSA] (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Potassium deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type II diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Unspecified nutritional deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Complete rupture of rotator cuff (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
"Degeneration of intervertebral disc, site unspecified" (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Degenerative joint disease (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Herniated disc (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leg pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar disc herniation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Shoulder bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of the prostate recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 2 (2)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast ductal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carcinoma hepatocellular (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Esophageal adenocarcinoma lower third in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Esophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 4 (4)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
"Malignant neoplasm of colon, unspecified" (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Oral carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 5 (7)
Renal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Renal clear cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma of the bladder stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign essential tremor (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 3 (4) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 2 (2) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic coma (Nervous system disorders) | 0 (0) | 1 (1)
Drug-induced encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Forehead headache (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (3)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 2 (2)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Myelitis transverse (Nervous system disorders) | 0 (0) | 1 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Oversedation (Nervous system disorders) | 1 (1) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Seizures (Nervous system disorders) | 0 (0) | 1 (1)
Simple partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 2 (2) | 2 (3)
Syncope (Nervous system disorders) | 3 (3) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1)
Upper motor neurone lesion (Nervous system disorders) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Addiction relapse (Psychiatric disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 5 (5)
Alcohol withdrawal syndrome (Psychiatric disorders) | 2 (2) | 0 (0)
Altercation (Psychiatric disorders) | 1 (1) | 0 (0)
Anger (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Attempted suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Auditory and visual hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
Auditory hallucinations (Psychiatric disorders) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 7 (7)
Depression worsened (Psychiatric disorders) | 0 (0) | 2 (2)
Dissociation (Psychiatric disorders) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 2 (3) | 1 (1)
Drug-induced psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 4 (6) | 6 (6)
Hypomania (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 3 (3) | 8 (8)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (2)
Opioid abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (2)
Polysubstance dependence (Psychiatric disorders) | 0 (0) | 1 (1)
Psychiatric disorder NOS (Psychiatric disorders) | 2 (2) | 0 (0)
Psychiatric symptom (Psychiatric disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic episode (Psychiatric disorders) | 0 (0) | 1 (1)
Stress symptoms (Psychiatric disorders) | 1 (1) | 1 (1)
Substance abuse (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal depression (Psychiatric disorders) | 2 (2) | 5 (6)
Suicidal ideation (Psychiatric disorders) | 29 (37) | 24 (37)
Suicidal plans (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 6 (9) | 2 (2)
Suicide gesture (Psychiatric disorders) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Kidney stones (Renal and urinary disorders) | 0 (0) | 2 (2)
Membranous nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteral calculus (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hypertrophy (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Enlarged prostate (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Ovarian cyst NOS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Aspiration pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthmatic attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Breath shortness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 5 (11) | 5 (6)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hilar mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Short of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Throat lesion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechial rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alcohol use (Social circumstances) | 1 (1) | 0 (0)
Burglary victim (Social circumstances) | 1 (1) | 0 (0)
Physical assault (Social circumstances) | 0 (0) | 1 (1)
Treatment noncompliance (Social circumstances) | 1 (1) | 0 (0)
Alcohol detoxification (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm repair (Surgical and medical procedures) | 1 (1) | 1 (1)
Appendectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Artificial urinary sphincter implant (Surgical and medical procedures) | 1 (1) | 0 (0)
Atherectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Back surgery (Surgical and medical procedures) | 0 (0) | 2 (2)
Bladder tumor resection (Surgical and medical procedures) | 1 (1) | 0 (0)
Bowel resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Bypass surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
C-section (Surgical and medical procedures) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Drug detoxification (Surgical and medical procedures) | 1 (1) | 0 (0)
Drug rehabilitation (Surgical and medical procedures) | 1 (1) | 0 (0)
Elective surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Foot surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Fusion cervical spine (Surgical and medical procedures) | 0 (0) | 1 (1)
Fusion of vertebra (Surgical and medical procedures) | 1 (1) | 0 (0)
Gallbladder operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastrostomy tube insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Hernia repair NOS (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip replacement (Surgical and medical procedures) | 0 (0) | 2 (2)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee operation (Surgical and medical procedures) | 1 (1) | 2 (2)
Knee total replacement (Surgical and medical procedures) | 1 (1) | 1 (1)
Lobectomy (thyroid) (Surgical and medical procedures) | 0 (0) | 1 (1)
Lumbar laminectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Lung operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Mass excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Penile operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Physical therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Prostate transurethral resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Rotator cuff repair (Surgical and medical procedures) | 0 (0) | 2 (2)
Shoulder replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Splenectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Total abdominal hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Total knee replacement (Surgical and medical procedures) | 2 (2) | 3 (3)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Uvulectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Wound drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Aneurysm of abdominal aorta (Vascular disorders) | 1 (1) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure high (Vascular disorders) | 2 (2) | 2 (2)
Deep vein thrombosis leg (Vascular disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotensive episode (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disease (Vascular disorders) | 2 (2) | 2 (2)
Peripheral vascular disease NOS (Vascular disorders) | 0 (0) | 1 (1)
Popliteal artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Superficial femoral arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Thrombosis arm (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis leg (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Integrated Care (N=472) | Standard of Care (N=471)
Unevaluable event (General disorders) | 2 (2) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Blurry vision (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gas (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upset stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 1 (1) | 1 (1)
Weight gain (Investigations) | 1 (1) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Abnormal thinking (Psychiatric disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Agitated (Psychiatric disorders) | 0 (0) | 1 (1)
Anger (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Auditory hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Bad dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Behavior abnormal (Psychiatric disorders) | 1 (1) | 1 (1)
Bizarre dreams (Psychiatric disorders) | 1 (1) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 4 (4)
Depression worsened (Psychiatric disorders) | 7 (7) | 3 (3)
Difficulty sleeping (Psychiatric disorders) | 2 (2) | 0 (0)
Dreaming excessive (Psychiatric disorders) | 0 (0) | 2 (2)
Emotional distress (Psychiatric disorders) | 1 (1) | 0 (0)
Frightening dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Increased agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Lack of motivation (Psychiatric disorders) | 0 (0) | 1 (1)
Mood change (Psychiatric disorders) | 2 (2) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Nightmares (Psychiatric disorders) | 2 (2) | 5 (5)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attacks (Psychiatric disorders) | 0 (0) | 1 (1)
Paranoia aggravated (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disturbance (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 6 (7) | 8 (8)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Violent behavior (Psychiatric disorders) | 1 (1) | 0 (0)
Vivid dreams (Psychiatric disorders) | 1 (1) | 3 (4)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Drug rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Generalized itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blood pressure high (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes